CLINICAL TRIAL: NCT07194109
Title: Remiazolam vs Propofol Total Intravenous Anesthesia on Postoperative Neurodevelopment After General Anesthesia in Children
Acronym: REMPPON
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PJ2025-06-90; 20250690 (Other: The First Affiliated Hospital of Anhui Medical University)
Record Dates: First submitted 2025-09-03; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-08

CONDITIONS: Adenotonsillar Hypertrophy
Keywords: remimazolam; neurodevelopment; propofol; children; tonsillectomy

STUDY DESIGN:
Intervention Model Description: randomized controlled clinical study
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam group (Experimental): patients who in this arm will receive remimazolam for general anesthesia induction and maintenance
  Interventions: Drug: Remimazolam based total intravenous anesthesia
- propofol group (Active Comparator): patients who in this arm will receive propofol for general anesthesia induction and maintenance
  Interventions: Drug: Propofol based general anesthesia

INTERVENTIONS:
Drug: Remimazolam based total intravenous anesthesia — For patients who aged between 3 and 6 years old undergoing tonsillectomy or/and adenoidectomy, anesthesia induction will performed with remimazolam in a dose of 0.4 - 0.5 mg/kg anesthesia maintenance was administered with remimazolam at a rate of 1.0 - 3.0 mg/kg/h.
  Arms: Remimazolam group
Drug: Propofol based general anesthesia — For patients who aged between 3 and 6 years old undergoing tonsillectomy or/and adenoidectomy, anesthesia induction will performed with propofol in a dose of 2.0 - 3.5 mg/kg , anesthesia maintenance was administered with propofol at a rate of 4 - 12 mg/kg/h.
  Arms: propofol group

SUMMARY:
The goal of this clinical trial is to learn the effects of remimazolam for total intravenous anesthesia on the neurodevelopment of children aged 3-6 years who underwent tonsil/adenoid removal surgery after general anesthesia when compared with propofol. It will also learn about the safety of remimazolam used for children. The main questions it aims to answer are:

* Does remimazolam improve the postoperative neurodevelopmental outcomes of the children after general anesthesia compared with propofol?
* What medical problems do participants have when receive remimazolam for general anesthesia? Researchers will compare remimazolam to propofol to see if remimazolam improve the postoperative neurodevelopmental outcomes of the children after general anesthesia.

Participants will:

* Receive remimazolam or propofol for general anesthesia induction and maintenance
* At 1-3 years after the surgery, the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition was used for face-to-face assessment of the children's neurodevelopmental status.
* Use scales such as BRIEF-P and CBCL to conduct face-to-face assessments of the patient's cognitive functions in other areas.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 3-6 years old;
2. Planned to undergo elective non-neurological, non-cardiac, and non-liver surgery under general anesthesia (abdominal surgery, orthopedic surgery, urological surgery, otolaryngological surgery, etc.);
3. Expected anesthesia duration to be more than 30 minutes;
4. ASA classification I-II;
5. BMI 14-25 kg/m2;
6. Postoperative plan not to be admitted to ICU;
7. Parents or legal guardians of the child have given informed consent;
8. Capable of communicating in Chinese.

Exclusion Criteria:

1. Those who were exposed to general anesthetic drugs during infancy or in the late pregnancy of the mother;
2. Known chromosomal abnormalities or other known acquired or congenital diseases that may affect neural development, such as cerebral palsy, autism spectrum disorder or attention deficit hyperactivity disorder (ADHD), etc.;
3. Patients with severe liver dysfunction (Child-Pugh C grade);
4. Patients with severe kidney dysfunction (requiring dialysis before surgery);
5. Patients with a history of congenital heart disease requiring surgery or drug treatment;
6. Those allergic to the study drugs remimazolam or propofol;
7. Any known neural damage, such as cystic periventricular leukomalacia or grade 3 or 4 intraventricular hemorrhage;
8. Social or geographical factors that may lead to postoperative loss of follow-up;
9. Planned to undergo two surgeries within 7 days after the surgery;
10. Those currently participating in other clinical trials;
11. Those receiving special care or living in social welfare institutions or any other factors that may affect their ability to participate in the study.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 558 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-10-01 (Estimated); Study Completion 2030-10-01 (Estimated)

PRIMARY OUTCOMES:
full-scale intelligence quotient | one year after surgery
  assessed by trained physicians, using the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (Chinese Version) 《WPPSI-IV(CN)》

SECONDARY OUTCOMES:
Memory and learning ability | The first to the third year after the operation
  assessed by trained physicians, using the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (Chinese Version) 《WPPSI-IV(CN)》
Language and Reading Skills | The first to the third year after the operation
  assessed by trained physicians, using the Wechsler Preschool and Primary Scale of Intelligence - Fourth Edition (Chinese Version) 《WPPSI-IV(CN)》
Executive Function and Attention | The first to third year after operation
  used by Behavior Rating Inventory of Executive Function for preschool (BRIEF-P)
Behavior and Emotion Assessment | The first to third year after surgery
  used by Achenbach Child Behavior Checklist (CBCL)
Motor development | The first to third years after surgery
  used by Movement Assessment Battery for Children-Second Edition(MABC-2)